CLINICAL TRIAL: NCT02539173
Title: Diagnosis of Diaphragmatic Paralysis After Interscalene Block by Measuring the Inspiratory Diaphragmatic Thickening: Feasibility and Impact Observed
Brief Title: Diagnosis of Diaphragmatic Paralysis After Interscalene Block: Feasibility and Impact Observed
Acronym: BBDDIAPHRAGM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FONCTION DIAPHRAGMATIQUE
Record Dates: First submitted 2015-08-26; First posted 2015-09-02 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2015-08

CONDITIONS: Shoulder Fractures; Arm Fractures
MeSH Terms: conditions — Shoulder Fractures | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): Ultrasound scan of diaphragm is made preoperatively during the pre-anesthetic visit, patients are informed of the purpose of the study. Written consent is collected after oral and written information.
  Interventions: Other: Ultrasound scan

INTERVENTIONS:
Other: Ultrasound scan — Non-invasive and non-irradiating. The diaphragmatic thickening in recovery is measured before and after the completion of the anesthetic block using the ultrasound system, the ultrasound probe and of an aqueous gel by trans-thoracic approach.
  It measures the thickness on deep inspiration and expiration in supine position. Each measurement is repeated twice. This measurement series lasts 4 minutes, is repeated 15 minutes after completion of the engine block when a block is found and contralateral. The total measurement time is about 12 minutes.

SUMMARY:
1. INTRODUCTION AND MAIN OBJECTIVES The incidence of diaphragmatic paralysis after an inter-block scalénique varies between 30 and 100% in the literature. Its clinical impact is mostly absent and paralysis regresses after the block lifted. When it is suspected, it can be diagnosed by a chest radio, showing an elevation of the dome.

   The objective of this study is to evaluate the incidence of diaphragmatic paralysis by measuring the thickness diaphragmatic as quantitative assessment of diaphragmatic contraction noninvasive ultrasound scan and feasibility of this measure in SSPI unit (post-interventional monitoring unit) with scan (ultrasound) in the usual way used for the block under ultrasound scan.
2. STUDY TYPE Prospective, single-center clinical study routine care involving 50 consecutive patients scheduled to undergo surgical procedures in the area of the shoulder or arm for which locoregional analgesia inter-block type scalénique or supraclavicular ultrasound scan is indicated below.
3. START OF THE STUDY February 2014 with an expected duration of six months.

DETAILED DESCRIPTION:
1. TITLE OF STUDY

   Diagnosis of diaphragmatic paralysis after interscalene block by measuring the inspiratory diaphragmatic thickening incidence and observed clinical consequences.
2. OBJECTIVES OF THE STUDY

   2.1 Primary Objective: To evaluate the incidence and clinical impact of diaphragmatic paralysis after interscalene block under ultrasound.

   To evaluate the clinical consequences of this paralysis. Quantify diaphragmatic paralysis: paralysis if present is it always complete.

   2.2 Secondary objective: Assess the feasibility of measuring the diaphragmatic thickening as a means simple diagnostics, rapid, non-invasive and non-irradiating bedside by the anesthetist in charge of the patient with the conventional ultrasound equipment available in the operating room without staff intervention Outdoor (radio manipulator, radiologist).
3. STUDY TYPE

   Single-center prospective study in routine care involving 50 consecutive patients conducted from February 2014 for 6 months.
4. LOCATION OF THE STUDY

   The study will take place in recovery and in the operating theater of the hospital Saint Joseph 185 Rue Raymond Losserand 75014 Paris.

   The information and the collection of patient consent will be held in pre-anesthetic visit.
5. RUNNING OF THE STUDY

5.1 Study Population Major patients scheduled to undergo surgical procedures in the area of the shoulder or arm for which locoregional analgesia inter-block type scalénique or supraclavicular ultrasound is indicated below.

5.2 anesthetic Protocol Block design: as recommended by SFAR, usual procedure In immediate preoperative patient monitored and infused, fractionated ultrasound-guided injection of 20 ml of 7.5% Naropin.

The surgery is then performed under general anesthesia according to the usual anesthetic protocol.

5.2 Recruitment Mode Preoperatively during the pre-anesthetic visit, patients are informed of the purpose of the study. Written consent is collected after oral and written information.

5.3 Data collection The collected data about the patient are ASA, weight, age, gender, block type, type of surgery, the occurrence of complications of the ALR, the administration of prophylactic antibiotics and dexamethasone , respiratory pathology history, renal function, drug class premedication, the occurrence of respiratory complications. The data is then entered in a EXCEL spreadsheet whose treatment will remain internal to GHPSJ.

5.4 Ultrasound examination of the diaphragm It is non-invasive and non-irradiating. The diaphragmatic thickening in recovery is measured before and after the completion of the anesthetic block using the ultrasound system, the ultrasound probe and of an aqueous gel by trans-thoracic approach.

It measures the thickness on deep inspiration and expiration in supine position. Each measurement is repeated twice. This measurement series lasts 4 minutes, is repeated 15 minutes after completion of the engine block when a block is found and contralateral. The total measurement time is about 12 minutes.

5.5 Diagnosis of diaphragmatic dysfunction Diaphragmatic paralysis is recognized when the inspiratory diaphragmatic thickening fraction is less than 20%.

7. SCHEDULED DATE FOR START OF THE STUDY: FEBRUARY 2014

9. PLANNED DURATION OF THE STUDY: 6 MONTHS

ELIGIBILITY:
Inclusion Criteria:

* Adults patients

Exclusion Criteria:

* Minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic thickening on deep inspiration and expiration in supine position. The fraction is estimated by percentage | The measurement series lasts 4 minutes, is repeated 15 minutes after completion of the engine block when a block is found and contralateral. The total measurement time is about 12 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Belaid BOUHEMAD, Dr, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France